CLINICAL TRIAL: NCT01560871
Title: Effects of a Walking Program and Inspiratory Muscle Training in Individuals With Chronic Heart Failure - A Pilot Study
Brief Title: Effects of a Walking Program and Inspiratory Muscle Training in Individuals With Chronic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Texas Health Resources (Other)
Responsible Party: Principal Investigator, Suh-Jen Lin, Associate Professor, Texas Woman's University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16969
Record Dates: First submitted 2012-03-20; First posted 2012-03-22 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Heart Failure NYHA Class II; Heart Failure NYHA Class III
Keywords: Heart failure; inspiratory muscle training; physical activity
MeSH Terms: conditions — Heart Failure; Motor Activity | interventions — Walking

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-intensity IMT Plus Walking (Sham Comparator): Inspiratory Muscle Training (IMT) intensity was set at 15% PImax. The walking program consisted of walking every day at an intensity of "somewhat hard" to "hard" on the Borg's Rating of Perceived Exertion (RPE) scale. Participants were encouraged to walk at 10 to 15 minutes, once to twice a day initially, then progressed to 45-50 minutes a day by the end of the six weeks, if they could tolerate.
  Interventions: Behavioral: Low-intensity IMT plus walking
- High-intensity IMT Plus Walking (Experimental): Inspiratory Muscle Training (IMT) intensity was set at 60% PImax.
  The walking program was the same as the one for the control group.
  Interventions: Behavioral: High-intensity IMT plus walking

INTERVENTIONS:
Behavioral: High-intensity IMT plus walking — The IMT intensity was set at 60% of PImax which was reassessed weekly. Frequency: 5x/week; 1x/day preferred. 6 Interval Levels: (6 efforts at each level): (1) 60s rest interval; (2) 45s rest interval; (3) 30s rest interval; (4) 15s rest interval; (5)10s rest interval; (6) 5s rest interval, trained to exhaustion.
  For the walking program, it was the same as the one for the control group.
  Arms: High-intensity IMT Plus Walking
Behavioral: Low-intensity IMT plus walking — The IMT training was 3 sets of 10 repetitions, or when the participant felt tired. Participants returned to our facility every week to reassess PImax.
  For the walking program, each participant was given a pedometer and a heart rate monitor to track daily step counts and heart rate. The walking program consisted of walking every day at an intensity of "somewhat hard" to "hard" on the Borg's Rating of Perceived Exertion scale. Participants began at least 10 to 15 minutes, once to twice a day, for 7 days a week, and eventually progressed to 45-50 minutes a day by the end of the six weeks, if they could tolerate.
  Arms: Low-intensity IMT Plus Walking

SUMMARY:
Individuals with chronic heart failure need a "safe and effective" exercise program that could enhance their quality of life. In this study, we examined whether an experimental exercise program of autonomous walking and high-intensity Inspiratory Muscle Training (IMT) could result in better effects on respiratory muscle strength (PImax), cardiovascular endurance, quality of life, and physical activity, when compared to autonomous walking and "sham" IMT program, in adults with chronic heart failure.

DETAILED DESCRIPTION:
Participants were recruited from the outpatient heart failure transitional care clinic at the Presbyterian Hospital of Dallas and other local heart failure support groups. Flyers were distributed to cardiologists, nurse practitioners, and local heart failure support groups in the Dallas/Ft Worth area. Cardiologists and nurse practitioners were aware of the scope of the study and its inclusion and exclusion criteria of research participants. Potential research participants could then call the research team for further information.

Participants came to our facility for the initial evaluation session, where a history interview was conducted to gather demographic data, such as age, gender, height, weight, race/ethnicity, and past medical/surgical history. The following baseline data were then collected: a) two trials of the six-minute walk test, b) respiratory muscle strength indicated by maximal inspiratory pressure (PImax), and two quality of life questionnaires. During the walk test, heart rate and heart rhythms were continuously monitored via a holter monitor. During the rest breaks, research participants filled out two quality of life questionnaires (SF-36, Minnesota Living with Heart Failure Questionnaire).

Each participant was randomly assigned to one of the two groups: a) the autonomous walking program with a high-intensity Inspiratory Muscle Training (IMT) program, or b) the autonomous walking program with a sham IMT. The training threshold for the experimental IMT group was trained at 60%PImax which was reassessed at weekly follow ups. The frequency of training was 5x/week (1x/day preferred) for 6 interval levels at each session (6 inspiratory efforts in each level): (1) 60s rest interval; (2) 45s rest interval; (3) 30s rest interval; (4) 15s rest interval; (5)10s rest interval; (6) 5s rest interval, trained to exhaustion. The intensity of sham IMT was set at fixed 15% PImax. Research participants were blinded to the group assignment. The time commitment for IMT was about 15-20 minutes a session per day at home. Weekly follow up was conducted at the School of Physical Therapy in Dallas to reassess PImax, collect the log of daily step count, and discuss about the walking program. Every participant was given a breathing device for inspiratory muscle training.

Each participant was given a pedometer and a heart rate monitor to track their daily step counts and heart rate during the walking session. The walking program consisted of walking daily at an intensity of "somewhat hard" to "hard" on the Borg's Rating of Perceived Exertion (RPE) scale. Participants were encouraged to walk 10 to 15 minutes, once to twice a day initially, then progressed to about 45-50 minutes a day by week six, if they could tolerate. At the end of 6 weeks, these participants returned to our facility for the final evaluation session.

ELIGIBILITY:
Inclusion Criteria:

* adults with chronic heart failure (NYHA Functional Class II-III)
* BMI < 35 kg/m^2
* Age: 18 to 90 years
* walk independently with or without an assisted device
* hospital discharge for CHF within a year.

Exclusion Criteria:

* ECG with uncontrolled ventricular arrhythmia
* bronchiectasis
* limited walking ability due to neurologic or orthopedic impairments of the legs

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-03; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Jen Lin, PhD, PT, Principal Investigator — Texas Woman's University
Locations (2):
- United States (2):
  - Outpatient heart failure transitional care clinic, Presbyterian Hospital of Dallas, Texas Health Resources, Dallas, Texas
  - School of Physical Therapy, Texas Woman's University, Dallas, Texas

REFERENCES:
- [Background] Gheorghiade M, Vaduganathan M, Fonarow GC, Bonow RO. Rehospitalization for heart failure: problems and perspectives. J Am Coll Cardiol. 2013 Jan 29;61(4):391-403. doi: 10.1016/j.jacc.2012.09.038. Epub 2012 Dec 5. PMID 23219302
- [Background] Van Spall HGC, Lee SF, Xie F, Oz UE, Perez R, Mitoff PR, Maingi M, Tjandrawidjaja MC, Heffernan M, Zia MI, Porepa L, Panju M, Thabane L, Graham ID, Haynes RB, Haughton D, Simek KD, Ko DT, Connolly SJ. Effect of Patient-Centered Transitional Care Services on Clinical Outcomes in Patients Hospitalized for Heart Failure: The PACT-HF Randomized Clinical Trial. JAMA. 2019 Feb 26;321(8):753-761. doi: 10.1001/jama.2019.0710. PMID 30806695
- [Background] Tudor-Locke C, Craig CL, Brown WJ, Clemes SA, De Cocker K, Giles-Corti B, Hatano Y, Inoue S, Matsudo SM, Mutrie N, Oppert JM, Rowe DA, Schmidt MD, Schofield GM, Spence JC, Teixeira PJ, Tully MA, Blair SN. How many steps/day are enough? For adults. Int J Behav Nutr Phys Act. 2011 Jul 28;8:79. doi: 10.1186/1479-5868-8-79. PMID 21798015
- [Background] Tudor-Locke C, Hart TL, Washington TL. Expected values for pedometer-determined physical activity in older populations. Int J Behav Nutr Phys Act. 2009 Aug 25;6:59. doi: 10.1186/1479-5868-6-59. PMID 19706192
- [Background] Bailly L, Mosse P, Diagana S, Fournier M, d'Arripe-Longueville F, Diagana O, Gal J, Grebet J, Moncada M, Domerego JJ, Radel R, Fabre R, Fuch A, Pradier C. "As du Coeur" study: a randomized controlled trial on quality of life impact and cost effectiveness of a physical activity program in patients with cardiovascular disease. BMC Cardiovasc Disord. 2018 Dec 6;18(1):225. doi: 10.1186/s12872-018-0973-3. PMID 30522438
- [Background] Lin SJ, McElfresh J, Hall B, Bloom R, Farrell K. Inspiratory muscle training in patients with heart failure: a systematic review. Cardiopulm Phys Ther J. 2012 Sep;23(3):29-36. PMID 22993500
- [Background] Marco E, Ramirez-Sarmiento AL, Coloma A, Sartor M, Comin-Colet J, Vila J, Enjuanes C, Bruguera J, Escalada F, Gea J, Orozco-Levi M. High-intensity vs. sham inspiratory muscle training in patients with chronic heart failure: a prospective randomized trial. Eur J Heart Fail. 2013 Aug;15(8):892-901. doi: 10.1093/eurjhf/hft035. Epub 2013 Mar 19. PMID 23512093
- [Background] Rector TS, Cohn JN. Assessment of patient outcome with the Minnesota Living with Heart Failure questionnaire: reliability and validity during a randomized, double-blind, placebo-controlled trial of pimobendan. Pimobendan Multicenter Research Group. Am Heart J. 1992 Oct;124(4):1017-25. doi: 10.1016/0002-8703(92)90986-6. PMID 1529875
- [Background] Middel B, Bouma J, de Jongste M, van Sonderen E, Niemeijer MG, Crijns H, van den Heuvel W. Psychometric properties of the Minnesota Living with Heart Failure Questionnaire (MLHF-Q). Clin Rehabil. 2001 Oct;15(5):489-500. doi: 10.1191/026921501680425216. PMID 11594639
- [Background] Neder JA, Andreoni S, Lerario MC, Nery LE. Reference values for lung function tests. II. Maximal respiratory pressures and voluntary ventilation. Braz J Med Biol Res. 1999 Jun;32(6):719-27. doi: 10.1590/s0100-879x1999000600007. PMID 10412550
- [Background] Borg GA. Psychophysical bases of perceived exertion. Med Sci Sports Exerc. 1982;14(5):377-81. PMID 7154893

RESULTS

PARTICIPANT FLOW:
Groups:
- Low-intensity IMT Plus Walking: Inspiratory Muscle Training (IMT) intensity is set at 15% PImax. The walking program consists of walking daily at an intensity of "somewhat hard" to "hard" on the Rating of Perceived Exertion scale. Participants are encouraged to walk 15 minutes twice a day, then progress to 45-50 minutes a day by six weeks.
  Low-intensity IMT plus walking: The IMT training is about 15-20 minutes. Both groups will need to come in once a week for 15 to 20 minutes to probably readjust the IMT training intensity on the breathing device.
  For the walking program, each participant will be given a pedometer and a heart rate monitor so he/she can track daily step counts and walking heart rate during the study. The walking program will consist of walking every day at an intensity of "hard" to "somewhat hard" on the Rating of Perceived Exertion (RPE) scale. Participants will begin walking at least 15 minutes twice a day for 7 days a week and eventually pr
- High-intensity IMT Plus Walking: Inspiratory Muscle Training (IMT) intensity is set at 60% PImax. The walking program will consist of walking daily at an intensity of "somewhat hard" to "hard" on the Rating of Perceived Exertion scale. Participants are encouraged to walk 15 minutes twice a day initially, then progress to 45-50 minutes a day by six weeks.
  High-intensity IMT plus walking: The IMT intensity will be set at 60% of PImax which will be adjusted weekly and nose clip will be used. Frequency: 5x/week; 1x/day preferred. 6 Interval Levels: (6 efforts at each level): (1) 60s rest interval; (2) 45s rest interval; (3) 30s rest interval; (4) 15s rest interval; (5)10s rest interval; (6) 5s rest interval, trained to exhaustion.
  For the walking program, each participant will be given a pedometer and a heart rate monitor so he/she can track daily step counts and heart rate during the study. The walking program will consist of walking every day at an intensity of "hard" to "somewhat har
Period: Overall Study
Arm/Group | Low-intensity IMT Plus Walking | High-intensity IMT Plus Walking
Started | 9 | 7
Completed | 3 | 5
Not Completed | 6 | 2
Not completed — transportation issues | 2 | 1
Not completed — relocation | 1 | 0
Not completed — readmission to a hospital | 2 | 1
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Low-intensity IMT Plus Walking: Inspiratory Muscle Training (IMT) intensity is set at 15% PImax. The walking program will consist of walking every day at an intensity of "hard" to "somewhat hard" on the Rating of Perceived Exertion (RPE) scale. Participants will be instructed to walk at 15 minutes twice a day initially, then progress to 45-50 minutes a day by the end of the six weeks.
  Low-intensity IMT plus walking: The IMT training is about 15-20 minutes. Both groups will need to come in once a week for 15 to 20 minutes to probably readjust the IMT training intensity on the breathing device.
  For the walking program, each participant will be given a pedometer and a heart rate monitor so he/she can track daily step counts and walking heart rate during the study. The walking program will consist of walking every day at an intensity of "hard" to "somewhat hard" on the Rating of Perceived Exertion (RPE) scale. Participants will begin walking at least 15 minutes twice a day for 7 days a week and eventually pr
- High-intensity IMT Plus Walking: Inspiratory Muscle Training (IMT) intensity is set at 60% PImax. The walking program will consist of walking every day at an intensity of "hard" to "somewhat hard" on the Rating of Perceived Exertion (RPE) scale. Participants will be instructed to walk 15 minutes twice a day initially, then progress to 45-50 minutes a day by the end of six weeks.
  High-intensity IMT plus walking: The IMT intensity will be set at 60% of PImax which will be adjusted weekly and nose clip will be used. Frequency: 5x/week; 1x/day preferred. 6 Interval Levels: (6 efforts at each level): (1) 60s rest interval; (2) 45s rest interval; (3) 30s rest interval; (4) 15s rest interval; (5)10s rest interval; (6) 5s rest interval, trained to exhaustion.
  For the walking program, each participant will be given a pedometer and a heart rate monitor so he/she can track daily step counts and heart rate during the study. The walking program will consist of walking every day at an intensity of "hard" to "somewhat har
- Total: Total of all reporting groups
Arm/Group | Low-intensity IMT Plus Walking | High-intensity IMT Plus Walking | Total
Number analyzed (Participants) | 9 | 7 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 6 | 6 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 6 | 15
  Unknown or Not Reported | 0 | 0 | 0
Six-Minute Walk Test Distance [Mean (Standard Deviation); unit: meters] — The six-minute walk test measures how far a person can walk in 6 minutes with his/her best effort. A longer distance indicates a better cardiovascular endurance.
  meters | 413.92 (85) | 356.00 (85.3) | 388 (109)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Minnesota Living With Heart Failure Questionnaire Score
Description: This questionnaire includes 21 questions which ask how much the heart condition affected the patient's life during the past month. Each question has 5 optional answers with the scores ranging from 0 to 5. A higher score indicates a worse outcome. The minimum overall score of the questionnaire is 0 and the maximum score is 105. A higher overall score on the Minnesota Living with Heart Failure Questionnaire indicates a worse outcome.
Time Frame: Baseline and 6 weeks
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Low-intensity IMT Plus Walking: For the low-intensity Inspiratory Muscle Training (IMT), the intensity was set at 15% maximal inspiratory pressure (PImax), which was considered "Sham training"..
  The walking program consisted of walking at an intensity of "hard" to "somewhat hard" on the Borg's Rating of Perceived Exertion scale. Participants were encouraged to walk at 15 minutes once to twice a day initially, then progress to a total of 45-50 minutes a day, if they could tolerate, by the end of six weeks. Every participant was given a pedometer and a polar heart rate monitor to track step counts and walking heart rate.
  The IMT training is about 15-20 minutes. Both groups came to our facility once a week for 15 to 20 minutes for discussions about their progress and readjustment of the training intensity on the IMT breathing device.
- High-intensity IMT Plus Walking: For the high-intensity Inspiratory Muscle Training (IMT), the intensity is set at 60% maximal inspiratory pressure (PImax). Frequency: 5x/week; 1x/day preferred. 6 rest Interval Levels: (6 efforts at each level): (1) 60s rest interval; (2) 45s rest interval; (3) 30s rest interval; (4) 15s rest interval; (5)10s rest interval; (6) 5s rest interval, trained to exhaustion.
  The walking program consisted of walking at an intensity of "hard" to "somewhat hard" on the Borg's Rating of Perceived Exertion scale. Participants were encouraged to walk at 15 minutes once to twice a day initially, then progress to a total of 45-50 minutes a day, if they could tolerate, by the end of six weeks. Every participant was given a pedometer and a polar heart rate monitor to track step counts and walking heart rate.
  Both groups returned once a week for discussions about their progress and readjustment of the IMT training intensity based on the new PImax measured..
Arm/Group | Low-intensity IMT Plus Walking | High-intensity IMT Plus Walking
Number analyzed (Participants) | 3 | 5
score on a scale
  MLHF score at baseline | 36 [11 to 66] | 57.6 [48 to 92]
  change from baseline at 6 weeks | 18.6 [-5 to 34] | -20.6 [-53 to 27]

2. Primary Outcome: Change From Baseline in Mean Score of Physical Component of the SF-36 Questionnaire
Description: The SF-36 quality of life questionnaire (short form) was used. A higher score of the SF-36 questionnaire indicates a better outcome (i.e., lower disability). The range of overall score on the SF-36 questionnaire is from 0 to 100.
Time Frame: Baseline and 6 weeks
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Low-intensity IMT Plus Walking | High-intensity IMT Plus Walking
Number analyzed (Participants) | 3 | 5
score on a scale
  Baseline Physical SF-36 | 34.1 [21.8 to 49.1] | 30.7 [23.4 to 40.4]
  Change from baseline physical SF-36 | 0.82 [-9.44 to 9.4] | 7.08 [2 to 17.6]

3. Secondary Outcome: Mean Daily Step Counts From Week 1 to Week 6
Description: Each subject was given a pedometer to record his/her step counts every day.
Time Frame: Baseline and 6 weeks
Measure: Mean (Full Range); unit: steps/day
Groups:
- High-intensity IMT Plus Walking: For the high-intensity Inspiratory Muscle Training (IMT), the intensity is set at 60% maximal inspiratory pressure (PImax). Frequency: 5x/week; 1x/day preferred. 6 rest Interval Levels: (6 efforts at each level): (1) 60s rest interval; (2) 45s rest interval; (3) 30s rest interval; (4) 15s rest interval; (5)10s rest interval; (6) 5s rest interval, trained to exhaustion.
  The walking program was the same as the one for the control group.
  Both groups returned once a week for discussions about their progress and readjustment of the IMT training intensity based on the new PImax measured..
Arm/Group | Low-intensity IMT Plus Walking | High-intensity IMT Plus Walking
Number analyzed (Participants) | 3 | 5
steps/day
  Baseline daily step count at Week 1 | 3512 [1051 to 6386] | 7002 [4222 to 9095]
  Daily step counts at week 6 | 4434 [1247 to 7798] | 9255 [4694 to 12173]

4. Secondary Outcome: Respiratory Muscle Strength is Indicated by Maximal Inspiratory Pressure (PImax)
Description: The inspiratory muscle strength will be measured in the unit of cmH2O by the Respiratory Muscle Pressure Meter (Micro Direct). A higher inspiratory pressure indicates a better inspiratory breathing strength.
Time Frame: Baseline and 6 weeks
Measure: Mean (Full Range); unit: cm H2O
Arm/Group | Low-intensity IMT Plus Walking | High-intensity IMT Plus Walking
Number analyzed (Participants) | 3 | 5
cm H2O
  Baseline PImax at week 1 | 51.44 [38 to 65] | 43.53 [19 to 72]
  PImax at week 6 | 57.22 [35.67 to 73.00] | 58.13 [38.00 to 81.00]

5. Secondary Outcome: Six-minute Walk Test Distance
Description: The six-minute walk test is a measure of cardiovascular endurance which measures how far a person can walk in 6 minutes. This test was conducted twice respectively at pre-training and at post-training to account for potential learning effect. A longer distance walked on the six-minute walking test indicates a better cardiovascular endurance.
Time Frame: Baseline and 6 Weeks
Measure: Mean (Full Range); unit: meters
Arm/Group | Low-intensity IMT Plus Walking | High-intensity IMT Plus Walking
Number analyzed (Participants) | 3 | 5
meters
  six-minute walk distance at week 1 | 356.16 [241.80 to 507.72] | 378.04 [353.57 to 415.26]
  Six-minute walk distance at week 6 | 375.78 [232.61 to 585.22] | 419.71 [365.46 to 465.73]

ADVERSE EVENTS:
Time Frame: Six weeks
Arm/Group | Low-intensity IMT Plus Walking | High-intensity IMT Plus Walking
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/7
Serious Adverse Events (participants affected / at risk) | 2/9 | 1/7
Other Adverse Events (participants affected / at risk) | 6/9 | 2/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-intensity IMT Plus Walking (N=9) | High-intensity IMT Plus Walking (N=7)
hospitalization (Cardiac disorders) | 0 (0) | 1 (1) — worsening of heart failure symptoms such as shortness of breath and weight gain.
hospitalization (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) — worsening of chronic obstructive pulmonary disease; pneumonia
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low-intensity IMT Plus Walking (N=9) | High-intensity IMT Plus Walking (N=7)
transportation issue, relocation, loss to follow up (Cardiac disorders) | 6 (6) | 2 (2) — Reasons for dropout: transportation issues (2), relocation (1), loss to follow up (1), hospital readmission (2 due to COPD or pneumonia)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-03-14): https://cdn.clinicaltrials.gov/large-docs/71/NCT01560871/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2013-12-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT01560871/Prot_SAP_001.pdf